CLINICAL TRIAL: NCT02865226
Title: Comparison of the Clinical Efficacy of 2 Paravertebral Block Strategies in Thoracic Surgery by Thoracotomy: : by the Anesthetist (Paravertebral Block Guided by Ultrasound) and by the Thoracic Surgeon (Paravertebral Block Visual)
Brief Title: Comparison of the Clinical Efficacy of 2 Paravertebral Block Strategies in Thoracic Surgery by Thoracotomy: by the Anesthetist (Paravertebral Block Guided by Ultrasound) and by the Thoracic Surgeon (Paravertebral Block Visual)
Acronym: PVBS-USguided
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA15082
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Pain
Keywords: thoracic surgery; thoracotomy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- experimental group (Experimental): paravertebral block by the anesthetist before incision (paravertebral block guided by ultrasound)
  Interventions: Other: paravertebral block by the anesthetist before incision (paravertebral block guided by ultrasound)
- control group (Active Comparator): paravertebral block by the thoracic surgeon at chest closure (paravertebral block visual)
  Interventions: Other: paravertebral block by the thoracic surgeon at chest closure (paravertebral block visual).

INTERVENTIONS:
Other: paravertebral block by the anesthetist before incision (paravertebral block guided by ultrasound)
  Arms: experimental group
Other: paravertebral block by the thoracic surgeon at chest closure (paravertebral block visual).
  Arms: control group

SUMMARY:
Post-thoracotomy pain is one of the most severe. The local analgesia allows its effective control and a reduction of postoperative morbidity and mortality.

The gold standard for local analgesia is the thoracic epidural. However, this technique can be dangerous with severe complications.

The paravertebral block showed comparable efficacy to the thoracic epidural for local analgesia . In addition, it has a better safety profile. There are several installation techniques. The difference in efficiency of these laying techniques is unknown.

DETAILED DESCRIPTION:
Compare the clinical effectiveness of two strategies of realization of paravertebral block: by the anesthetist before incision (paravertebral block guided by ultrasound) and by the thoracic surgeon at chest closure (paravertebral block visual).

ELIGIBILITY:
Inclusion Criteria:

* patient with thoracotomy indication for segmentectomy (s), lobectomy (s) lung or pulmonary wedge resection
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

* patient with neuropathy
* patient with body mass index superior to 35 kg/m2
* patient with contraindication for paravertebral block or local analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
pain | 24 hours
  Pain evaluated using a visual analog pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France